CLINICAL TRIAL: NCT01789697
Title: Using Mobile Phone Text Messaging and E-mailing to Decrease Anxiety, Pain, Follow-up Visits and Improve Reporting of Surgical Site Infection After Spine Surgery: A Double-Blind Randomized Trial
Brief Title: Text Message Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not sufficient staff to complete the trial.
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00034182
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Anxiety; Pain; Surgical Site Infection
MeSH Terms: conditions — Anxiety Disorders; Pain; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Receives text messages/emails (Experimental): Will receive text messages and emails periodically from the surgeon from Day 1 (day after discharge) through day 21.
  Interventions: Other: cellular device/computers
- Does not receive text messages/emails (No Intervention): Will not receive text messages and emails periodically from the surgeon from Day 1 (day after discharge) through day 21.

INTERVENTIONS:
Other: cellular device/computers — A random group of patients will receive text messages to their cellular device from the surgeon, as well as emails to their email addresses.
  Arms: Receives text messages/emails

SUMMARY:
The objectives of this double-blind, randomized, controlled study are to evaluate the efficacy of maintaining contact with low-back pain patients through text messaging and emailing, to decrease anxiety levels, pain, number of follow-up visits through text messaging and emailing, and to improve reporting of surgical site infection after spine surgery through text messaging and emailing. The outcomes that will be measured are anxiety, pain, follow-up visits and received phone calls, and reporting signs of surgical site infection. Participants will include Dr. Oren Gottfried's patients who underwent spine surgery at Duke Hospital or at Duke Raleigh Hospital. Patients will be approached after determination that the patient is going to undergo spinal surgery. All patients meeting inclusion criteria will be approached to participate irrespective of race or ethnicity. A total of 194 subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Patients age greater than 18 years
* Patients who confirm they have an unlimited text message data plan and email capabilities on their mobile device
* Patients of Dr. Gottfried's underwent lumbar decompression or fusion surgery
* Patients with text message capabilities
* Patients who have an active email account

Exclusion Criteria:

* Patients who demonstrate an inability to fill out the pre-visit questionnaires
* Patients with a diagnosis of metastatic disease
* Patients with workers compensation or liability pending
* Patients who will require transfer to an acute rehabilitation facility following surgery

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-09; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Change in Anxiety | Day 1-21, Month 3, Month 12
  Anxiety is measured by the Zung Self-Rating Anxiety Scale, which will be filled out everyday from day 1 (day after discharge) through day 21, and at the 3 month and 12 month mark.
Change in Pain | Day 1-21, Month 3, Month 12
  Pain is measured by the VAS Scale, which will be filled out everyday from day 1 (day after discharge) through day 21, and at the 3 month and 12 month mark.
Change in Surgical Site | Day 1-21
  Changes in the surgical site is measured by a questionnaire, which will be filled out everyday from day 1 (day after discharge) through day 21.

CONTACTS AND LOCATIONS:
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States